CLINICAL TRIAL: NCT02833168
Title: Validation of a German Language Screening Questionnaire for Symptoms of Respiratory Muscle Weakness and Sleep-disordered Breathing in Patients With Neuromuscular Disorders
Brief Title: Screening Questionnaire for Respiratory Muscle Weakness and Sleep-disordered Breathing in Neuromuscular Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universität Münster (Other)
Responsible Party: Principal Investigator, Matthias Boentert, MD, Senior Consultant in Neurology and Sleep Medicine, Universität Münster
Other Study IDs: KSN_2016_1_MB
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Neuromuscular Disorders
Keywords: Neuromuscular disorders; Sleep disordered breathing; Dyspnea
MeSH Terms: conditions — Neuromuscular Diseases; Sleep Apnea Syndromes; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients with proven neuromuscular disorders known to be potentially associated with significant diaphragmatic weakness, e. g. ALS, myotonic dystrophy type 1, limb-girdle muscular dystrophy, Duchenne and Becker muscular dystrophy. Patients already receiving home ventilatory support will not be included in the study.
  Interventions: Other: patient-filled questionnaires; Device: spiromanometry
- 2: Patient with proven obstructive sleep apnea syndrome prior to CPAP initiation.
  Interventions: Other: patient-filled questionnaires; Device: spiromanometry
- 3: Patients with sleep disorders other than sleep-related breathing disorders, e. g. narcolepsy, hypersomnia, parasomnia or sleep-related movement disorders.
  Interventions: Other: patient-filled questionnaires; Device: spiromanometry

INTERVENTIONS:
Other: patient-filled questionnaires — All patients answer selected questionnaires on sleep-related symptoms, sleep quality, daytime performance, and health-related quality of life.
Device: spiromanometry — Measurement of forced vital capacity, maximum inspiratory pressure and maximum expiratory pressure

SUMMARY:
It is the aim of this project to develop and validate a German language screening questionnaire for symptoms of respiratory muscle weakness and sleep-disordered breathing (SDB) in patients with neuromuscular disorders.

DETAILED DESCRIPTION:
SDB is a promiment clinical feature of various neuromuscular disorders including amyotrophic lateral sclerosis (ALS), spinal muscular atrophy (SMA), and myopathies such as myotonic dystrophy type 1, Pompe disease, and limb-girdle muscular dystrophies (LGMD). In ALS, SMA, LGMD and Pompe disease, SDB is usually caused by nocturnal alveolar hypoventilaton due to diaphragmatic weakness which manifests first during sleep and REM sleep in particular. SDB usually leads to sleep disruption, non-restorative sleep and daytime symptoms including morning headache, hypersomnolence, and increased neuromuscular fatigue. In patients with severe diaphragmatic involvement both symptoms of SDB and potential complications of respiratory muscle weakness substantially add to overall disease burden of the disease and decrease life span. Diagnosis of SDB is established by means of sleep studies which should ideally comprise polysomnography (PSG) and transcutaneous capnography. PSG with capnometry is time-consuming, expensive and not readily available for patients or referring physicians, respectively. For this reason it is desirable to thoroughly screen patients with neuromuscular disease for symptoms of SDB and respiratory muscle weakness. Results from a validated screening questionnaire could be used as an adjunctive to pulmonary function testing or spirometry results in order to identify patients in whom sleep studies should be performed. In addition, a screening questionnaire would facilitate early recognition of patients with SDB, enabling treating physicians to take appropriate steps to establish the diagnosis and to initiate non-invasive ventilation as early as possible.

Until now, there is no validated German language screening questionnaire for symptoms of respiratory muscle weakness and SDB. Steier et al. published an English language questionnaire which was validated as a screening tool in 33 patients with very different neuromuscular disorders which were predominantly neurogenic (Steier et al. 2011). In this study, SDB was defined by an apnea hypopnea index above 5 per hour. Nocturnal oxygen saturation and CO2 monitoring were not taken into account at all. In addition the questionnaire does not systematically cover sleep-related symptoms of SDB in detail (such as sleep disruption and morning headache) which have to be separated from daytime symptoms such as dyspnea or orthopnea, respectively.

Thus, the current project aims to correlate comprehensively generated items of a screening questionnaire with sleep study results including capnography alongside with respiratory muscle testing in patients with neuromuscular disorders. As control subjects, patients with newly diagnosed obstructive sleep apnea syndrome and sleep disorders other than sleep-related breathing disorders are enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* proven neuromuscular disease known to be potentially associated with diaphragmatic weakness (group 1)
* newly diagnosed obstructive sleep apnea with an apnea hypopnea index > 15/h total sleep time (group 2)
* newly diagnosed narcolepsy, hypersomnia, insomnia or parasomnia in the absence of any sleep-related breathing disorder (group 3)
* availability of recent diagnostic sleep studies including polysomnography and transcutaneous capnography

Exclusion Criteria:

* ongoing CPAP oder non-invasive ventilation
* inability to participate in study procedures
* severe lung disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuromuscular disorders, newly diagnosed obstructive sleep apnea syndrome or sleep disorders other than sleep-related breathing disorders (30 patients in each group)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Nocturnal hypercapnia tcCO2 | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Boentert, MD, Study Chair — University Hospital Münster, Department of Sleep Medicine and Neuromuscular Disorders
Locations (2):
- Germany (2):
  - University Hospital Münster, Department of Sleep Medicine and Neuromuscular Disorders, Münster
  - Bethanien Hospital, Solingen